CLINICAL TRIAL: NCT04604067
Title: Assessing a Circulating Tumor (ctDNA) and Positron Emission Tomography (PET)-Oriented Therapy in Patients With Diffuse Large B-cell Lymphoma (DLBCL). A Multicenter, Open-label, Phase II Trial.
Brief Title: Assessing a ctDNA and PET-oriented Therapy in Patients With DLBCL A Multicenter, Open-label, Phase II Trial.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 38/19; 2020-003876-42 (EudraCT Number)
Record Dates: First submitted 2020-10-22; First posted 2020-10-27 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Diffuse large B-cell lymphoma; Circulating tumor DNA (ctDNA); PET-oriented therapy; acalabrutinib-R-CHOP; acalabrutinib
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — acalabrutinib

STUDY DESIGN:
Intervention Model Description: All patients will have a PET/CT (PET1) and evaluation of circulating tumor DNA (ctDNA1) at baseline. The trial consists of four treatment cohorts (cohorts A, B, C and D) and a first assignment to treatment will be done at baseline based on the presence or absence of MYD88 L265P and/or CD79A/B mutations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm with 4 cohorts (Experimental): Cohort A: MYD88 L265P and/or CD79A/B mutations at baseline Treatment: Acalabrutinib-R-CHOP for a total number of 6 cycles.
  Cohort B, C D: Without MYD88 L265P and CD79A/B mutations at baseline:
  Assignment of cohort B, C and D after 2 cycles of R-CHOP according to PET (Deauville score (DS)) and molecular response (MR) (>2log10 reduction of ctDNA) results:
  Cohort B: DS 4 and No MR Treatment: 2 cycles of acalabrutinib-R-CHOP. After PET3/ctDNA3: patients with DS 1-3 and no MR OR DS4 with MR will receive 2 additional cycles of acalabrutinb-R-CHOP and 2 cycles of acalabrutinib single agent.
  Cohort C: DS 1-3 and MR Treatment: 2 additional cycles of R-CHOP (4x RCHOP in total) followed by 2 cycles of rituximab single agent.
  Cohort D: DS 4 and no MR OR DS 1-3 and MR Treatment: 4 additional cycles of RCHOP (6 cycles in total).
  Follow up: Patients off treatment will be followed for 5 years.
  Interventions: Drug: Acalabrutinib

INTERVENTIONS:
Drug: Acalabrutinib — Cohort A: 6 cycles of acalabrutinib-R-CHOP
  Cohort B: 2 cycles of R-CHOP and 2 cycles of acalabrutinb-R-CHOP followed by 2 cycles of acalabrutinib single agent
  Cohort C: 4 cycles of R-CHOP followed by 2 cycles of rituximab single agent
  Cohort D: 6 cycles of R-CHOP
  Rituximab 375 mg/m2 IV Day 1, cyclophosphamide 750 mg/m2 IV Day 1, doxorubicin 50 mg/m2 IV Day 1, vincristine 1.4 mg/m2 (maximum 2 mg) IV Day 1; prednisone 100 mg PO d1-5; Acalabrutinib 100 mg BID Day 1-21, cycles repeated every 21 days

SUMMARY:
Within this exploratory multicohort phase II trial, SAKK aims to evaluate a PET/CT and ctDNA oriented therapy in DLBCL in order to test the following working hypothesis.

* acalabrutinib-R-CHOP may improve the progression free survival in genetically defined DLBCL harboring the MYD88 L265P and/or CD79A/B mutations;
* treatment escalation to acalabrutinib-R-CHOP in DLBCL patients who have positive PET/CT (with residual disease scored as Deauville score 4 or 5 with centrally defined response) and no molecular response (<2log10 reduction of ctDNA) after two courses of R-CHOP could improve the anti-tumour activity of R-CHOP;
* treatment de-escalation to 4 total R-CHOP courses plus 2 rituximab single agent infusions does not compromise the outcome in patients lacking both MYD88 L265P and CD79A/B mutations and quickly obtaining both negative PET/CT (Deauville score 1-3) and molecular response (>2log10 reduction of ctDNA) after two cycles of R-CHOP.

DETAILED DESCRIPTION:
Despite advances in the clinical care of patients with DLBCL and in understanding the biology of this disease, cure rates have remained the same since the introduction of rituximab to CHOP chemotherapy, and R-CHOP chemoimmunotherapy remains the standard of care. Over the last years many phase III trials investigating new agents added to R-CHOP have been performed but they have all invariably failed to improve treatment outcomes. Importantly, three of the most recently completed phase III trials that were developed based on the cell of origin distinction of DLBCL and aimed to improve treatment outcome in the ABC (or non- Germinal center B-Cell (GCB)) subtype by adding a targeted agent to R-CHOP have also failed. This provides clinical evidence that cell of origin may not be an accurate biomarker for treatment decisions. The R - CHOP + investigational drug approach has thus failed either when broadly applied to unselected DLBCL patients or when applied to DLBCL patients selected according to inaccurate biomarkers such as COO.

Within this exploratory multicohort phase II trial, SAKK aims to evaluate a PET/CT and ctDNA oriented therapy in DLBCL in order to test the following working hypothesis.

* acalabrutinib-R-CHOP may improve the progression free survival in genetically defined DLBCL harboring the MYD88 L265P and/or CD79A/B mutations;
* treatment escalation to acalabrutinib-R-CHOP in DLBCL patients who have positive PET/CT (with residual disease scored as Deauville score 4 or 5 with centrally defined response) and no molecular response (<2log10 reduction of ctDNA) after two courses of R-CHOP could improve the anti-tumour activity of R-CHOP;
* treatment de-escalation to 4 total R-CHOP courses plus 2 rituximab single agent infusions does not compromise the outcome in patients lacking both MYD88 L265P and CD79A/B mutations and quickly obtaining both negative PET/CT (Deauville score 1-3) and molecular response (>2log10 reduction of ctDNA) after two courses R-CHOP.

Primary objectives:

* Assessing the efficacy of acalabrutinib-R-CHOP in DLBCL harboring MYD88 L265P and/or CD79A/B mutations (cohort A)
* Assessing the activity of treatment escalation to acalabrutinib-R-CHOP followed by acalabrutinib monotherapy in DLBCL patients who are double positive: PET/CT positive (Deauville score 4 or 5 with centrally defined response) and no molecular response (<2log10 fold reduction) after two courses of R-CHOP (cohort B)
* Exploring the feasibility of treatment de-escalation to 4 total R-CHOP courses plus two infusions of single agent rituximab in patients lacking both MYD88 L265P and CD79A/B mutations and quickly obtaining both negative PET/CT (Deauville score 1-3) and molecular response (>2log10 reduction of ctDNA) after two cycles of R-CHOP (cohort C).
* Exploring clinical implications of having a negative PET/CT (Deauville score 1-3) but no molecular response (<2log10 reduction of ctDNA) vs a positive PET/CT (Deauville score 4 or 5 with centrally defined response) but molecular response (>2log10 reduction of ctDNA) after two R-CHOP courses (cohort D)

Secondary objectives:

* Safety and tolerability of acalabrutinib-R-CHOP
* Assessment of prognostic value of baseline PET radiomics indexes, alone or in association with other parameters

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to ICH GCP E6(R2) regulations before registration and prior to any trial specific procedures.
* Histologically confirmed, treatment-naïve DLBCL, NOS that fulfill all the following:
* Patient eligible for 6 cycles of R-CHOP
* Ann Arbor stage I-IV
* Metabolically active measurable disease by 18FDG PET-CT
* No previous treatment with systemic chemotherapy or radiotherapy (a pre-phase treatment with steroids for up to a total of 10 days is allowed; baseline PET/CT, liquid biopsy and bone marrow biopsy and aspirate must be collected either before or within a maximum of 5 days after steroid pre-phase treatment starts. If a patient receives steroids, glucose levels must be checked and be normal on the day of PET/CT before the exam.
* At least 1 measurable site of disease according to Revised Response Criteria for Malignant Lymphoma. The site of disease must be greater than 1.5 cm in the long axis regardless of short axis measurement or greater than 1.0 cm in the short axis regardless of long axis measurement, and clearly measurable in 2 perpendicular dimensions.
* Quantifiable and qualifiable circulating tumor DNA
* Patients with a prior malignancy and treated with curative intention are eligible if all treatment of that malignancy was completed at least 2 years before registration and the patient has no evidence of disease at registration. Less than 2 years is acceptable for malignancies with low risk of recurrence and/or no late recurrence.
* Age ≥ 18 years
* EGOG performance status 0-2 (or 3 if due to disease)
* Adequate bone marrow function: neutrophil count ≥ 1.0 x 109/L, platelet count ≥ 75 x 109/L (unless due to bone marrow involvement: in this case the permitted limit is ≥ 50 x 109/L) with allowed premedication or supportive medication.
* Adequate hepatic function: total bilirubin ≤ 1.5 x ULN (except for patients with Gilbert's disease ≤ 3.0 x ULN), AST, ALT ≤ 2.5 x ULN, or ≤ 5 x ULN under the assumption that abnormal values are a result of liver involvement by lymphoma
* Adequate renal function: estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73 m2 (according to CKD-EPI formula)
* Adequate cardiac function: Left ventricular Ejection Fraction (LVEF) ≥ 50% as determined by echocardiography (ECHO)
* Adequate coagulation function: INR ≤ 1.5 x ULN (the ULN for INR is defined with the value 1.2 for all sites, in case no ULN is documented in the lab certificates/sheets), aPTT ≤ 1.5 x ULN.
* Women of childbearing potential must use highly effective contraception, are not pregnant or lactating and agree not to become pregnant during trial treatment and until 12 months after the last dose of investigational drug. A negative pregnancy test before inclusion into the trial is required for all women of childbearing potential. (www.swissmedicinfo.ch).
* Men agree not to donate sperm or to father a child during trial treatment and until 12 months after the last dose of investigational drug
* Patient is able and willing to swallow trial drug as whole capsule or tablet.
* Patient is willing to participate in translational research projects

Exclusion criteria:

* CNS lymphoma involvement
* Stage I disease that has been completely surgically excised (not measurable)
* Specific diagnostic categories of large B-cell lymphoma such as high grade B-cell lymphoma, primary mediastinal large B-cell lymphoma, primary central nervous system lymphoma, T-cell/histiocyte-rich large B-cell lymphoma, intravascular large B-cell lymphoma, plasmablastic lymphoma, lymphomatoid granulomatosis, primary effusion lymphoma or transformed lymphoma etc.
* Concomitant treatment with any other experimental drug
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV; unstable angina pectoris, history of myocardial infarction within the last six months, serious arrhythmias requiring medication (with exception of asymptomatic or rate controlled atrial fibrillation or paroxysmal supraventricular tachycardia), significant QT-prolongation, uncontrolled hypertension.
* Uncontrolled systemic infection.
* History of or ongoing confirmed progressive multifocal leukoencephalopathy (PML).
* History of cerebrovascular accident or intracranial hemorrhage within 6 months prior to registration
* History of bleeding diathesis (eg, haemophilia, von Willebrand disease).
* Major surgery in the preceding 4 weeks of first dose of study drug. If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of the stomach or small bowel, gastric bypass, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction or gastric restrictions and bariatric surgery, such as gastric bypass.
* History or presence of clinically relevant central nervous system (CNS) pathology as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis.
* Known history of human immunodeficiency virus (HIV) or active chronic hepatitis C or hepatitis B virus infection or any uncontrolled active systemic infection requiring intravenous (iv) antimicrobial treatment. All patients must be screened for HIV up to 28 days prior to study drug start using a blood test for HIV according to local regulations. All patients must be screened for hepatitis up to 28 days prior to study drug start using the routine hepatitis virus laboratory panel. Patients positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) will be eligible if they are negative for HBV-DNA, these patients should receive prophylactic antiviral therapy and have HBV-DNA testing every 4 months. Patients positive for anti-HCV antibody will be eligible if they are negative for HCV-RNA.
* Active, uncontrolled autoimmune phenomenon (autoimmune hemolytic anemia or immune thrombocytopenia) requiring steroid therapy with > 20 mg daily of prednisone dose or equivalent.
* Requires or receiving anticoagulation with warfarin or equivalent antagonists (eg, phenprocoumon), 'dual' antiplatelet therapy (DAPT), such as aspirin and clopidogrel. However, use of therapeutic low molecule weight heparin, direct oral anticoagulants, or low dose anti-platelet agents is allowed.
* Concomitant treatment to acalabrutinib capsules or tablets with strong CYP3A inducers or strong CYP3A inhibitors. The use of strong CYP3A inhibitors within 1 week or strong CYP3A inducers within 3 weeks of the first dose of acalabrutinib is prohibited.
* Co-administration of acalabrutinib capsules with proton pump inhibitors (PPIs).
* Any concomitant drugs contraindicated for use with the trial drugs according to the approved product information
* Known hypersensitivity to trial drug(s) or to any component of the trial drug(s)
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-06-25 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Cohorts A, C and D: Progression free survival (PFS) according to the Lugano criteria | from registration until the first event as defined in PFS (estimated 2 years)
  PFS is defined as the time from registration until the first event of interest:
  * Progressive disease according to the Lugano Classification
  * Death from any cause
  Patients not having an event at the time of analysis and patients starting a new anticancer therapy in the absence of an event will be censored at the date of their last tumor assessment showing non-progression before starting a new treatment.
Cohort B: Complete remission (CR) rate at the end of therapy according to the Lugano criteria | estimated 9 months after registration
  Patients with CR at the end of therapy will be considered CR. Patients with no tumor assessment at the end of therapy will be considered:
  * non-CR, if they have no following tumor assessment within the trial (patient died, refused, started a new treatment or was lost to follow-up) or if they have non-CR at the following tumor assessment after the end of therapy.
  * CR, if they have CR at the following tumor assessment after end of therapy before starting a new treatment.

SECONDARY OUTCOMES:
Adverse events (AEs) | record throughout treatment phase (until 28 days after last dose of trial treatment)
  All AEs will be assessed according to NCI CTCAE v5.0.
Overall survival (OS) | from registration to date of death from any cause (estimated 5 years)
  OS will be calculated from registration until death from any cause. Patients not experiencing an event will be censored at the last date they were known to be alive.
Progression free survival in cohort B | from registration until the first event as defined in PFS (estimated 2 years)
  Analogous to the evaluation of the primary endpoint of cohorts A, C and D, but in cohort B.
Complete remission rate in cohorts A, C and D | estimated 9 months after registration
  Analogous to the evaluation of the primary endpoint of cohort B, but in cohorts A, C and D.
Overall response rate (ORR) | estimated 9 months after registration
  ORR at the end of therapy is defined as either PR or CR (OR) according to the Lugano criteria. Patients with no tumor assessment at the end of therapy will be considered:
  * non-OR, if they have no following tumor assessment within the trial (patient died, refused, started a new treatment or was lost to follow-up) or if they have non-OR at the following tumor assessment after the end of therapy.
  * OR, if they have OR at the following tumor assessment after end of therapy before starting a new treatment
Duration of response (DoR) | estimated 2 years
  The DoR will be calculated from when the criteria for CR or PR are met, until documentation of progressive disease thereafter. Only patients with a CR or PR will be included in this analysis. Patients without any documentation of progressive disease thereafter will be censored at the last date of tumor assessment without progression and before the start of a new anti-lymphoma treatment, if any.

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios Stathis, Prof, Study Chair — IOSI, Ospedale San Giovanni Bellinzona
Locations (19):
- Italy (3):
  - Ospedale Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera Universitaria Maggiore della Carita di Novara, Novara
  - Policlinico Agostino Gemelli, Roma
- Switzerland (16):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden (Baden/Brugg), Baden
  - St. Claraspital, Basel
  - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Inselspital, Bern, Bern
  - Kantonsspital Graubünden, Chur
  - Hopital Fribourgeois, Fribourg
  - Hopitaux Universitaire de Genève (HUG), Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Luzern, Luzerne
  - Réseau Hospitalier Neuchâtelois (RHNe), Neuchâtel
  - Kantonsspital Olten, Olten
  - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - UniversitätsSpital Zürich, Zurich
  - City Hospital Triemli, Zurich